CLINICAL TRIAL: NCT02991287
Title: Prospective External Validation of a Predictive Scale of Chronic Postsurgical Pain
Brief Title: Validation of Predictive Scale of Chronic Postsurgical Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Antonio Montes, Anesthesiologyst, PhD., Parc de Salut Mar
Other Study IDs: PI16/00279
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hysterectomy, Vaginal; Thoracotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic post-surgical pain patients: Patients scheduled for differents types of surgery (inguinal, hernia repair, abdominal hysterectomy, vaginal hysterectomy, and thoracotomy).
  Interventions: Procedure: Inguinal hernia repair; Procedure: Abdominal hysterectomy; Procedure: Vaginal hysterectomy; Procedure: Thoracotomy

INTERVENTIONS:
Procedure: Inguinal hernia repair
Procedure: Abdominal hysterectomy
Procedure: Vaginal hysterectomy
Procedure: Thoracotomy

SUMMARY:
To asses the precision of a score to predict chronic post surgical pain in patients undergoing inguinal hernia repair, abdominal hysterectomy, vaginal hysterectomy and thoracotomy. Prospective multicenter cohort study in 21 hospital in spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with given inform consent, aged mor than 18 years, who undergo scheduled surgery of one of the following types: inguinal hernia (men), abdominal hysterectomy, vaginal hysterectomy and thoracotomy (men)

Exclusion Criteria:

* Patients aged less than 18 years,
* Patients requiring reoperation because of surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All spanish patients who undergo scheduled surgery of one of the following types:
  inguinal herniorrhaphy, abdominal hysterectomy, vaginal hysterectomy, thoracotomy.
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Estimated)
Dates: Start 2017-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
GENDOLCAT scale punctuations (composed by 6 items: type of surgery, age, pain in area of surgery, pain in other localisations, physical component of SF12 and mental component of SF12). | After evaluation of chronic postsurgical pain 4th month after the end of surgery
  GENDOLCAT scale punctuations (composed by 6 items: type of surgery, age, pain in area of surgery, pain in other localisations, physical component of SF12 and mental component of SF12) to identify patients that could develop chronic post surgical pain after inguinal hernia repair, abdominal hysterectomy, vaginal hysterectomy and thoracotomy.

SECONDARY OUTCOMES:
Verbal rating scale | After evaluation of chronic postsurgical pain 4th month after the end of surgery
  Prevalence of chronic post surgical pain after inguinal hernia repair, abdominal hysterectomy, vaginal hysterectomy and thoracotomy will be assessed by verbal rating scale.

CONTACTS AND LOCATIONS:
Locations (21):
- Spain (21):
  - Hospital de Badalona, Badalona, Barcelona
  - Hospital Germans Tries i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital de la Vall d'Hebrón, Barcelona, Barcelona
  - Hospital de Sant Rafael, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital de Cruces, Barakaldo, Bizcaia
  - Hospital de Galdakao, Bizkaia, Bizkaia
  - Hopsital Gregorio Marañon, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Son Espases, Palma de Mallorca, Palma
  - Hospital Son Llatzer, Palma de Mallorca, Palma
  - Hospital Nuestra Señora de Valme, Seville, Sevilla
  - Hospital General de Alicante, Alicante, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Lluís Alcanyís de Xàtiva, Valencia, Valencia
  - Hospital de Valladolid, Valladolid, Valladolid

REFERENCES:
- [Derived] Montes A, Roca G, Cantillo J, Sabate S; GENDOLCAT Study Group. Presurgical risk model for chronic postsurgical pain based on 6 clinical predictors: a prospective external validation. Pain. 2020 Nov;161(11):2611-2618. doi: 10.1097/j.pain.0000000000001945. PMID 32541391